CLINICAL TRIAL: NCT03914963
Title: Efficacy of a Fibrin Sealant (Tissucol Duo®) for the Prevention of Lymphocele After Laparoscopic Pelvic Lymphadenectomy Due to Gynaecological Cancer: a Randomised Controlled Trial
Brief Title: Efficacy of a Fibrin Sealant for the Prevention of Lymphocele After Lymphadenectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IBON JAUNARENA (Other)
Responsible Party: Sponsor-Investigator, IBON JAUNARENA, Gynecologist Oncologist, Hospital Donostia
Organization: Hospital Donostia (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ONC-1111
Record Dates: First submitted 2018-08-16; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lymphocele
Keywords: Fibrin Tissue Adhesive; Lymph node dissection
MeSH Terms: conditions — Lymphocele

STUDY DESIGN:
Intervention Model Description: After standard preoperative assessment, patients were randomly assigned to having Tissucol Duo® applied to the surgical bed in only the right or only the left hemipelvis after bilateral pelvic lymphadenectomy. Following the manufacturer´s instructions, 5 ml of sealant was sprayed evenly across the entire surgical bed in only one hemipelvis (the treated hemipelvis). We decided to treat only one hemipelvis in each patient, thereby allowing patients to serve as their own controls, in order to compare outcomes with and without the sealant in the same body with the same clinical characteristics and reduce the influence of other factors beyond the treatment.
Who Masked: Outcomes Assessor
Masking Description: The patient, doctors who performed the follow-up and initially the surgeon were blinded to the randomization sequence and site of application. That is, the surgeon was only told to which hemipelvis the sealant was to be applied when he considered that the surgical procedure had been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fibrin sealant treatment hemipelvis (Experimental): •Drug: Following the manufacturer´s instructions, 5 ml of sealant was sprayed evenly across the entire surgical bed in only one hemipelvis (the treated hemipelvis).
  Interventions: Biological: Fibrin sealant hemipelvis
- Control hemipelvis (Placebo Comparator): Other hemipelvis
  Interventions: Biological: Control hemipelvis

INTERVENTIONS:
Biological: Fibrin sealant hemipelvis — Following the manufacturer´s instructions, 5 ml of sealant was sprayed evenly across the entire surgical bed in only one hemipelvis (the treated hemipelvis) after pelvis bilateral lymphadenectomy.
  Arms: Fibrin sealant treatment hemipelvis
Biological: Control hemipelvis — Contralateral hemipelvis not treated with fibrin sealant
  Arms: Control hemipelvis

SUMMARY:
Objective:

Lymphocele (LC) is a potential complication of lymph node removal. The objective of this study was to assess the efficacy of the Tissucol Duo® (Baxter AG Industriestrasse 67 A-1221 Vienna, Austria) fibrin sealant in decreasing the incidence of LC after pelvic laparoscopic lymph node dissection using harmonic shears.

Material and Methods:

This prospective double blind randomised study was conducted between February 2012 and June 2016 in Donostia University Hospital (Spain). Overall, 74 patients diagnosed with gynaecological cancer gave written informed consent and were included in the study. After bilateral pelvic lymphadenectomy, the fibrin sealant was used following manufacturer's instructions in one hemipelvis but not the other. Overall, the product was applied in 41 (55.4%) left and 33 (44.6%) right hemipelvises. The primary objective of the study was to determine the incidence of LC after surgery in symptomatic and asymptomatic patients. Imaging (ultrasound, computed tomography and magnetic resonance) was performed to detect LC at 3, 6 and 12 months after surgery.

DETAILED DESCRIPTION:
This prospective double blind randomized study was conducted by the Gynaecological Cancer Unit of Donostia University Hospital (San Sebastian, Basque Country, Spain) between February 2012 and June 2016. The study was approved on 24 August 2012 by the clinical research ethics committee of our hospital (study reference number ONC-1111).

All patients diagnosed with gynaecological (cervical, endometrial or ovarian) cancer due to undergo transperitoneal bilateral laparoscopic pelvic lymphadenectomy (LPL) as part of their surgical treatment were invited to participate. Our treatment protocol is based on clinical guidelines of the European Society Gynaecology and Oncology and the Spanish Society of Gynaecology and Obstetrics (SEGO).

The inclusion criteria were that the patient had endometrial, cervical, or ovarian cancer, underwent PL, an expected survival of more than 12 weeks and appropriate bone marrow, kidney and liver function, as well as that they agreed to participate and signed the informed consent form. Patients were excluded if they had previously received radiotherapy or chemotherapy, haematological disorders including coagulation defects, a history of thromboembolic disease or lymphatic system disorders (lymphedema or lymphocele), or allergy to aprotinin, as well as if they declined to participate or did not sign the informed consent form.

After standard preoperative assessment, patients were randomly assigned to having Tissucol Duo® applied to the surgical bed in only the right or only the left hemipelvis after bilateral LPL. The patient, doctors who performed the follow-up and initially the surgeon were blinded to the randomization sequence and site of application. That is, the surgeon was only told to which hemipelvis the sealant was to be applied when he considered that the surgical procedure had been completed. Following the manufacturer´s instructions, 5 ml of sealant was sprayed evenly across the entire surgical bed in only one hemipelvis (the treated hemipelvis). Using this protocol, the investigators sought to minimise intervention bias, in that the surgeon did not know where he was going to spray the sealant until the end of the LPL procedure. The investigators decided to treat only one hemipelvis in each patient, thereby allowing patients to serve as their own controls, in order to compare outcomes with and without the sealant in the same body with the same clinical characteristics and reduce the influence of other factors beyond the treatment.

All the patients received antithrombotic and antibiotic prophylaxis according to our usual protocols and were operated on by the same surgical team, all procedures being carried out using ultrasonic shears (Harmonic®, Ethicon, Cincinnati, OH, USA) In patients with endometrial cancer, we also carried out retroperitoneal aortocaval lymphadenectomy as part of surgical staging (para-aortic lymph node dissection PALND, as described by Querleu) up to the left renal vein, followed by type A radical hysterectomy (Querleu-Morrow 2011/EORT) and opening of the retroperitoneal space after the surgical intervention. In patients with cervical cancer, after LPL and intraoperative lymph node biopsy, the surgeons completed surgery with transperitoneal aortic lymphadenectomy if the biopsy was positive or radical hysterectomy (type B1 or C1) if it was negative.

The limits of the dissection of the LPL were: the psoas muscle laterally, the obliterated umbilical artery medially, the crossing of the ureter over the common iliac artery cranially, and the crossing of the circumflex iliac vein over the external iliac artery caudally. The caudal limit of the aortocaval dissection was the bifurcation of the aorta, with the cranial limit being the level of both renal veins, and all lymphatic tissue was removed from the paracaval, interaortocaval, paraaortic and presacral regions between the ureters.

Data were collected on the following variables: age, body weight, height, type of tumour, tumour stage (FIGO), surgical procedure, duration of surgery, intra and postoperative complications, length of hospital stay, readmission, and number of lymph nodes obtained in each area, as well as the presence, location, size and symptoms of LCs and changes over time in these parameters.

Routine follow-up assessments conducted at 3, 6 and 12 months after surgery included imaging, ultrasound, computed tomography or magnetic resonance, depending on which was indicated for monitoring the patient's cancer. The imaging findings were used to assess the incidence of LC, defined as the accumulation of lymphatic fluid, in particular along the iliac vessels, the observer for this examination being blind to patient group allocation. These follow-up findings were compared to imaging (ultrasound, computed tomography or magnetic resonance) results prior to the surgery.

The sample size was calculated assuming an overall incidence of LC after LPL of 30%, based on previous studies. The investigators estimated that a sample of at least 39 hemipelvises for each study arm was needed to declare a 34% (Tinelli et al) lower incidence of LC with the treatment as significant with an alpha of 0.05 and beta of 0.1.

All the patient clinical and surgical data were entered into a Microsoft Access 2010 database. Once cleaned, data were imported into IBM SPSS Statistics for Windows, version 21.0 (Armonk, NY, USA) for statistical analysis. Data were summarised using the mean and standard deviation for quantitative variables and absolute and relative frequencies expressed as percentages for qualitative variables.

The analysis was performed per protocol. To assess the efficacy of the intervention, chi-square or Fisher's exact tests were used to compare the rate of LC in the two groups (intervention and control), while Student's t test for unpaired samples was used to compare parametric variables between groups. Significance was set at a value of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient had endometrial, cervical, or ovarian cancer, underwent PL, an expected survival of more than 12 weeks and appropriate bone marrow, kidney and liver function, as well as that they agreed to participate and signed the informed consent form

Exclusion Criteria:

* Patients were excluded if they had previously received radiotherapy or chemotherapy, haematological disorders including coagulation defects, a history of thromboembolic disease or lymphatic system disorders (lymphedema or lymphocele), or allergy to aprotinin, as well as if they declined to participate or did not sign the informed consent form.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
assess the efficacy of the Tissucol Duo® (Baxter AG Industriestrasse 67 A-1221 Vienna, Austria) fibrin sealant in decreasing the incidence of LC after pelvic laparoscopic lymph node dissection using harmonic shears | 12 months
  Tissucol Duo®, marketed under the name of Tisseel® Fibrin Sealant in some countries, is a physiological haemostatic sealant containing fibrinogen and thrombin with haemostatic, sealant, adhesive and healing properties. It can be employed in laparoscopic surgery using a spray system that that spreads the product across the wound surface and, in theory, can help to seal lymph vessels and thereby reduce the incidence of lymphadenectomy and associated complications. The objective of this prospective study was to assess the efficacy of Tissucol Duo® sealant in decreasing the incidence of LC after laparoscopic pelvic lymphadenectomy using harmonic shears

CONTACTS AND LOCATIONS:
Overall Officials: IBON JAUNARENA, Consultant, Principal Investigator — Hospital Donostia

IPD SHARING:
Plan to Share IPD: Undecided